CLINICAL TRIAL: NCT00778778
Title: Blinded, Comparative, Randomized, Single-Dose, Three Way Crossover Bioavailability Study of Ranbaxy and Bristol-Myers Squibb Company (CEFZIL ®) 500 mg Cefprozil Tablets in Healthy Adult Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Cefprozil Tablets, USP 500 mg Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: AA27168
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence cefprozil 500mg tablets fasting conditions
MeSH Terms: interventions — Cefprozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Cefprozil 500mg tablets of ranbaxy
  Interventions: Drug: cefprozil 500mg tablets
- 2 (Active Comparator): CEFZIL ® 500 mg cefprozil tablets of BMS, USA
  Interventions: Drug: cefprozil 500mg tablets
- 3 (Active Comparator): CEFZIL ® 500 mg tablets, BMS Canada
  Interventions: Drug: cefprozil 500mg tablets

INTERVENTIONS:
Drug: cefprozil 500mg tablets

SUMMARY:
The objective of this study was to assess the single-dose relative bioavailability of Ranbaxy and Bristol-Myers Squibb Company (CEFZIL ®) 500 mg cefprozil tablets, under fasting conditions.

DETAILED DESCRIPTION:
This was a blinded, randomized, single dose, 3-way crossover comparative bioavailability study performed on 27 healthy adult volunteers (13 males and 14 females). In each period, subjects were housed from at least 10 hours before dosing until after the 10 hour post dose events. Subjects received a single oral 500 mg cefprozil dose of their assigned formulation, with 240 mL of water under fasting condition. Food was restricted from 10 hours before dosing until 4 hours post dose and water was not permitted from 2 hours before dosing and was restricted until 2 hours following dosing but was allowed ad libitum at all other times. The doses were separated by a washout period of 14 days.

A total of twenty seven (27) healthy adult volunteers (13 males and 14 females) were enrolled in the study, out of which only twenty four (24) subjects (11 males and 13 females) completed the clinical phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject candidates fulfilled all of the following inclusion criteria to be eligible for the participation in the study, unless otherwise specified.

  1. Healthy adult male or female volunteers, 18 - 55 years of age;
  2. Weighing at least 52 kg for males and 45 kg for females and within 15% of their ideal weights (Table of " Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983);
  3. Medically healthy subjects with clinically normal laboratory profiles, vital signs and ECGs.
  4. Females of childbearing potential were to be either sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or using one of the following acceptable birth control methods:
* surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum;
* IUD in place for at least 3 months;
* Barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study;
* Surgical sterilization of the partner (vasectomy for 6 months minimum);
* Hormonal contraceptives for at least 3 months prior to the first dose of the study
* Other birth control methods may have been deemed acceptable e) Postmenopausal women with amenorrhea for at least 2 years were eligible f) Voluntarily consented to participate in the study

Exclusion Criteria:

* Subjects were excluded from the study if there was evidence of any of the following at screening or at any time during the study:

  1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
  2. In addition, history or presence of :
* alcoholism or drug abuse within the past year;
* hypersensitivity or idiosyncratic reaction to cefprozil, other cephalosporin antibiotics, or penicillin;
* Female subjects who were pregnant or lactating. c) Positive results on HIV, HbsAg and/ or HCV tests. d) Subjects who were on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study e) Subjects who through completion of the study, would have donated in excess of:
* 500 mL of blood in 14 days, or
* 1500 mL of blood in 180 days, or
* 2500 mL of blood in 1 year. f) Subjects who participated in another clinical trial within 28 days prior to the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2005-05; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Saint-Laurent, Montreal, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html